CLINICAL TRIAL: NCT04836702
Title: Vascular Surgery Outcomes: Echocardiography as Risk-Assessment for Major Adverse Cardiac Events in Major Vascular Surgery Patients
Brief Title: Echocardiography as Risk-Assessment for Major Adverse Cardiac Events in Major Vascular Surgery Patients
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Margaret Clarke Tracci, Principal Investigator, University of Virginia
Other Study IDs: 20906
Record Dates: First submitted 2021-04-01; First posted 2021-04-08 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Left-Sided Heart Failure; Right-Sided Heart Failure; Heart Valve Diseases
Keywords: major vascular surgery; major adverse cardiac events
MeSH Terms: conditions — Heart Failure; Heart Valve Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Left ventricular function: * Depressed LV function
    1. LV ejection fraction < 50%
    2. LV systolic function; defined as mild / mod / sev decreased
    3. LV diastolic function; defined as mild (g1 ) / mod (g2) / sev ( g3) decreased
  * Normal LV function
- Right ventricular function: * Depressed RV function
    a. RV systolic function defined as mild / mod / sev decreased
  * Normal RV function
- Valvular lesions: * Moderate or severe valvular lesions
    1. Aortic stenosis
    2. Aortic regurgitation
    3. Mitral stenosis
    4. Mitral regurgitation
    5. Tricuspid regurgitation
  * Clinically normal valvular lesions
    1. No valvular lesion
    2. Mild stenosis / regurgitation of above mentioned lesions

SUMMARY:
Patient with coronary artery disease (CAD), heart failure and abnormal heart function undergoing major vascular surgery have a high associated high morbidity and mortality with myocardial infarction accounting for 33-50% of perioperative deaths. The prevalence of CAD in vascular surgery patients approaches 50%. Proper pre-procedure protocols to accurately assess patients and determine who may require further medical optimization prior to undergoing surgery help mitigate risk and improve outcomes. The investigators designed this study as a single center, retrospective cohort analysis to explore the association between ventricular (LV and RV function) and valvular (Aortic / Mitral / Tricuspid) function and expanded major adverse cardiac events (X-MACE).

ELIGIBILITY:
Inclusion Criteria:

* Major vascular surgery operation (e.g. CEA, open aortic repair, suprainguinal and infrainguinal bypasses, EVAR, TEVAR) captured in the UVA Vascular Quality Initiative database
* Echocardiography within two years of index operation

Exclusion Criteria:

* If patient had additional qualifying vascular procedure within 30 days of the index operation, this procedure was excluded

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent major vascular surgery operations at the University of Virginia
Sampling Method: Non-Probability Sample
Enrollment: 813 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Expanded Major Adverse Cardiac Events | In-hospital admission (within 120 days of index surgery)
  Composite outcome defined as any cardiovascular death, non-fatal MI, non-fatal stroke, post-operative CHF, or new dysrhythmias, all within the index hospital admission.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Meyer, MD, Study Director — Assistant Professor of Anesthesiology at University of Virginia

IPD SHARING:
Plan to Share IPD: Undecided
Will be made on an individual basis in accordance with guidance from the IRB and VQI panel

REFERENCES:
- [Background] Reis PV, Lopes AI, Leite D, Moreira J, Mendes L, Ferraz S, Amaral T, Mourao J, Abelha F. Major Cardiac Events in Patients Admitted to Intensive Care After Vascular Noncardiac Surgery: A Retrospective Cohort. Semin Cardiothorac Vasc Anesth. 2019 Sep;23(3):293-299. doi: 10.1177/1089253218825442. Epub 2019 Jan 25. PMID 30678531
- [Background] Golubovic M, Peric V, Stanojevic D, Lazarevic M, Jovanovic N, Ilic N, Djordjevic M, Kostic T, Milic D. Potential New Approaches in Predicting Adverse Cardiac Events One Month after Major Vascular Surgery. Med Princ Pract. 2019;28(1):63-69. doi: 10.1159/000495079. Epub 2018 Nov 4. PMID 30391950
- [Background] Ouriel K, Green RM, DeWeese JA, Varon ME. Outpatient echocardiography as a predictor of perioperative cardiac morbidity after peripheral vascular surgical procedures. J Vasc Surg. 1995 Dec;22(6):671-7; discussion 678-9. doi: 10.1016/s0741-5214(95)70057-9. PMID 8523601
- [Background] Flu WJ, van Kuijk JP, Hoeks SE, Kuiper R, Schouten O, Goei D, Elhendy A, Verhagen HJ, Thomson IR, Bax JJ, Fleisher LA, Poldermans D. Prognostic implications of asymptomatic left ventricular dysfunction in patients undergoing vascular surgery. Anesthesiology. 2010 Jun;112(6):1316-24. doi: 10.1097/ALN.0b013e3181da89ca. PMID 20502115
- [Background] Lerman BJ, Popat RA, Assimes TL, Heidenreich PA, Wren SM. Association of Left Ventricular Ejection Fraction and Symptoms With Mortality After Elective Noncardiac Surgery Among Patients With Heart Failure. JAMA. 2019 Feb 12;321(6):572-579. doi: 10.1001/jama.2019.0156. PMID 30747965
- [Background] Matyal R, Hess PE, Subramaniam B, Mitchell J, Panzica PJ, Pomposelli F, Mahmood F. Perioperative diastolic dysfunction during vascular surgery and its association with postoperative outcome. J Vasc Surg. 2009 Jul;50(1):70-6. doi: 10.1016/j.jvs.2008.12.032. PMID 19563954
- [Derived] Meyer MJ, Jameson SA, Gillig EJ, Aggarwal A, Ratcliffe SJ, Baldwin M, Singh KE, Clouse WD, Blank RS. Clinical implications of preoperative echocardiographic findings on cardiovascular outcomes following vascular surgery: An observational trial. PLoS One. 2023 Jan 19;18(1):e0280531. doi: 10.1371/journal.pone.0280531. eCollection 2023. PMID 36656845

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT04836702/Prot_SAP_001.pdf